CLINICAL TRIAL: NCT05238493
Title: A Phase 1, Randomized, Double Blind, Placebo Controlled, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VEL-101 Administered Intravenously or Subcutaneously in Healthy Subjects.
Brief Title: A Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VEL-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: VEL-101.KI102
Record Dates: First submitted 2022-01-25; First posted 2022-02-14 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Subcutaneous (SQ) Dose "A" (Experimental): Single dose of VEL-101 by SQ injection
  Interventions: Drug: VEL-101
- Intravenous (IV) Dose "A" (Experimental): Single dose of VEL-101 by IV infusion
  Interventions: Drug: VEL-101
- SQ Dose "B" (Experimental): Single dose of VEL-101 by SQ injection
  Interventions: Drug: VEL-101
- SQ Dose "C" (Experimental): Single dose of VEL-101 by SQ injection
  Interventions: Drug: VEL-101
- IV Dose "C" (Experimental): Single dose of VEL-101 by IV infusion
  Interventions: Drug: VEL-101
- SQ Dose "D" (Experimental): Single dose of VEL-101 by SQ injection
  Interventions: Drug: VEL-101
- SQ Dose "E" (Experimental): Single dose of VEL-101 by SQ injection
  Interventions: Drug: VEL-101
- SQ or IV Placebo (Placebo Comparator): Single dose of Placebo by SQ injection or IV infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VEL-101 — Intervention administered via subcutaneous injection or 1-hour intravenous infusion on Day 1
  Arms: IV Dose "C"; Intravenous (IV) Dose "A"; SQ Dose "B"; SQ Dose "C"; SQ Dose "D"; SQ Dose "E"; Subcutaneous (SQ) Dose "A"
Drug: Placebo — Intervention administered via subcutaneous injection or 1-hour intravenous infusion on Day 1
  Arms: SQ or IV Placebo

SUMMARY:
This study is primarily designed to assess the safety and tolerability of single doses of VEL-101 when administered subcutaneously (via injection into an area under the skin) or intravenously (via infusion into a vein). As each new group of participants is enrolled into the study, the dose administered to that group may be higher than a previous dose shown to be safe in other participants. The study is also designed to determine blood levels of VEL-101 and some substances produced by the immune system following VEL-101 administration. This information can provide insight into how quickly VEL-101 is eliminated from the body and some if its effects on the body.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the key components of the study as described in the written informed consent document, and willing and able to provide written informed consent;
2. Self-described healthy male or female, 18 to 65 years of age, inclusive, at Screening;
3. Body mass index (BMI) within the range of 18.5 to <35 kg/m2 at Screening;
4. If female, is surgically sterile, 2 years postmenopausal, or, if of childbearing potential, is using a medically accepted method of contraception (abstinence, the simultaneous use of 2 barrier methods, or the use of an intrauterine device [in place at least 3 months prior to dosing], or oral contraceptives), and agrees to continued use of this method until study Day 50;
5. If male, agrees to use an approved method of contraception (abstinence, 2 barrier methods, female partner's use of an intrauterine device [in place at least 3 months prior to dosing], oral contraceptives or female partner who is surgically sterile or 2 years postmenopausal) and agrees to use this method until study Day 50;
6. Able to comply with all study procedures, including the required overnight stays in the clinical research center and the food, beverage, and medication restrictions during the study;
7. In the opinion of the Investigator, is able to adhere to the requirements of the study.

Exclusion Criteria:

1. Known allergy to study medication or its components (non-medicinal ingredients) or a history of a severe allergic reaction to any drug or history of multiple food/drug allergies;
2. Use of tobacco, smoking cessation products, or products containing nicotine within 3 months prior to Screening;
3. History of alcohol or illicit drug use disorder, marijuana consumption as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th edition, or a reported habitual alcohol intake greater than 1.5 oz (ethanol equivalent) per day (eg, 24 oz of beer, 10 oz of wine, or 3 oz of hard liquor) for the past two years;
4. Positive urine screen for drugs of abuse including tetrahydrocannabinol or has a positive breathalyzer test on admission to the study center, at Screening and at Baseline for each treatment cohort;
5. Positive serologic test for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV), or positive for EBV polymerase chain reaction [PCR] at Screening;
6. Negative for Epstein-Barr Virus ([EBV], viral capsid antigen [VCA IgG], Epstein-Barr nuclear antigen antibody [EBNA],);
7. History of inadequately treated active or latent mycobacterium tuberculosis (TB) infection or positive QuantiFERON® TB Gold at Screening;
8. History of diabetes, clinically significant cardiovascular, pulmonary, hepatic, renal, or malabsorptive disease, as determined by the Principal Investigator (PI);
9. Clinically significant abnormality upon physical examination at Screening, as determined by the Investigator;
10. Clinically significant abnormality on 12-lead ECG at Screening, as determined by the Investigator;
11. Clinically significant abnormal laboratory values (clinical chemistry, hematology, coagulation, or urinalysis) outside the reference values established by the laboratory, as determined by the Investigator at Screening;
12. Positive pregnancy test or lactating at Screening or at Day -1;
13. Participation in an investigational study within 30 days or within 5 half-lives of the investigational drug, whichever is longer, prior to the Screening Visit;
14. Receiving any antibody or biologic medicinal product within 90 days prior to Screening;
15. Blood or plasma donation within 72 hours prior to Screening or planned up to study Day 50;
16. Positive test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) antigen testing or equivalent testing on Day -1; Subjects fully recovered from coronavirus disease 2019 (COVID-19) infection are eligible. Subjects with a past history of hospitalization due to COVID-19 infection will be excluded;
17. History of infection or vaccination within 90 days prior to the Screening, or planned vaccination within 90 days of dosing, with the exception of vaccination against SARS CoV-2;
18. History or presence, upon clinical evaluation, of any illness that, in the opinion of the Investigator, would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the subject at undue risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Number and Percentage of Participants with Treatment-emergent Adverse Events (TEAEs) | Day 1 through Day 50
  Number and percentage of participants experiencing one or more adverse events which occurred or worsened in severity after initiation of investigational product (IP) dosing
Number and Percentage of Participants with Serious TEAEs | Day 1 through Day 50
  Number and percentage of participants experiencing one or more serious TEAEs
Number and Percentage of Participants with Grade 3 or Higher TEAEs | Day 1 through Day 50
  Number and percentage of participants experiencing one or more grade 3 TEAEs
Number and Percentage of Participants with TEAEs Leading to Withdrawal from the Study | Day 1 through Day 50
  Number of participants experiencing one or more TEAEs directly resulting in withdrawal from the study
Number and Percentage of Participants with TEAEs Leading to Death | Day 1 through Day 50
  Number and percentage of participants experiencing TEAEs that resulted in death

SECONDARY OUTCOMES:
Number and Percentage of Participants with Abnormal Chemistry Panel Results | Days -1, 2 (24 hours), 3, 5, 8, 15, 22, 29, 50
  Descriptive statistics will summarize results (including change from baseline, as appropriate) of the following at each time point: sodium, potassium, chloride, calcium, bicarbonate, glucose, phosphorus, blood urea nitrogen, creatinine, creatine kinase, C-reactive protein, estimated glomerular filtration rate (eGFR), magnesium, amylase, uric acid, alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transferase (GGT), albumin, alkaline phosphatase, direct bilirubin, total bilirubin, indirect bilirubin, total protein, and lactate dehydrogenase
Number and Percentage of Participants with Abnormal Hematology Panel Results | Days -1, 2 (24 hours), 3, 5, 8, 15, 22, 29, 50
  Descriptive statistics will summarize results (including change from baseline, as appropriate) of the following at each time point: hematocrit, hemoglobin, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW), red blood cells (RBC), white blood cells (WBC) and differential, and platelets
Number and Percentage of Participants with Abnormal Coagulation Panel Results | Days -1, 2 (24 hours), 3, 5, 8, 15, 22, 29, 50
  Descriptive statistics will summarize results (including change from baseline, as appropriate) of the following at each time point: prothrombin time (PT), international normalized ratio (INR), partial thromboplastin time (PTT), and fibrinogen
Number and Percentage of Participants with Abnormal Urinalysis Results | Days -1, 2 (24 hours), 3, 5, 8, 15, 22, 29, 50
  Descriptive statistics will summarize results (including change from baseline, as appropriate) of the following at each time point: specific gravity, pH, leukocytes, erythrocytes, protein, glucose, nitrite, urobilinogen, bilirubin, ketones, and additional microscopic examination if blood or protein are abnormal
Number and Percentage of Participants with Abnormal 12-lead Electrocardiogram (ECG) Results | Days 1 (0, 1, 2, 3, 4, 5, 8, 12, 12, 16, and 20 hours), 2 (24, 30, 36, and 42 hours), 3, 4, 5, 8, 29, 50
  Descriptive statistics will summarize results (including change from baseline, as appropriate) of the following at each time point: PR interval, QRS duration, QT interval, corrected QT interval (QTc), and corrected QT interval using Fridericia's formula (QTcF)
Number and Percentage of Participants with Abnormal Vital Signs Results | Days -1, 1 (0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 8, 12, 16, 20 hours), 2 (24, 30, 36, 42 hours), 3, 4, 5, 6, 7, 8, 15, 22, 29, 50
  Descriptive statistics will summarize results (including change from baseline, as appropriate) of the following at each time point: heart rate (HR), respiratory rate (RR), blood pressure (BP), temperature, and oxygen saturation
CD28 Receptor Occupancy | Day 1 (0, 1, 3, 5, 8 hours) and Days 2 (24 hours), 3, 15, 22, 29, 50
  Proportion of target receptors occupied by VEL-101
Number and Percentage of Participants with Anti-drug Antibody (ADA) Formation | Days 1 (0 hour), 15, 29, 50
  Presence of detectable anti-VEL-101 antibodies; neutralizing antibody assessments to be performed in samples positive for ADA
Number and Percentage of Participants with Detectable Systemic Cytokine Concentrations | Day 1 (0, 1, 3, 5, 8 hours) and Days 2 (24 hours), 3, 15, 50
  Interferon-gamma, interleukin-1 beta, interleukin-2, interleukin-4, interleukin-5, interleukin-6, interleukin-8, interleukin-10, interleukin-13, interleukin-17, interleukin-12 p70 (heterodimer composed of p40 and p35 subunits), tumor necrosis factor-alpha
Maximum Plasma Concentration (Cmax) | Day 1 (0, 1, 3, 5, 8 hours) and Days 2 (24 hours), 3, 4, 5, 6, 7, 8, 15, 22, 29, 50
  The observed maximum plasma concentration
Time of Observed Maximum Plasma Concentration (Tmax) | Day 1 (0, 1, 3, 5, 8 hours) and Days 2 (24 hours), 3, 4, 5, 6, 7, 8, 15, 22, 29, 50
  Time at which the observed maximum plasma concentration occurred
Terminal Elimination Rate Constant | Day 1 (0, 1, 3, 5, 8 hours) and Days 2 (24 hours), 3, 4, 5, 6, 7, 8, 15, 22, 29, 50
  Terminal elimination rate constant, determined using the linear least squares regression of the terminal phase of the log plasma concentration time profile
Terminal Elimination Half-life | Day 1 (0, 1, 3, 5, 8 hours) and Days 2 (24 hours), 3, 4, 5, 6, 7, 8, 15, 22, 29, 50
  Elimination half-life calculated using terminal phase plasma concentration data
Area Under the Plasma Concentration Versus Time Curve (AUC) from Time Zero to Time of Last Observed Quantifiable Concentration | Day 1 (0, 1, 3, 5, 8 hours) and Days 2 (24 hours), 3, 4, 5, 6, 7, 8, 15, 22, 29, 50
  Area under the plasma concentration versus time curve (AUC) from time zero to time of last observed quantifiable concentration (different from AUC from time zero to infinity)
AUC from Time Zero to Infinity | Day 1 (0, 1, 3, 5, 8 hours) and Days 2 (24 hours), 3, 4, 5, 6, 7, 8, 15, 22, 29, 50
  Area under the plasma concentration versus time curve from time zero to infinity
Total Clearance (CL) | Day 1 (0, 1, 3, 5, 8 hours) and Days 2 (24 hours), 3, 4, 5, 6, 7, 8, 15, 22, 29, 50
  Total clearance from plasma
Terminal Volume of Distribution (Vz) | Day 1 (0, 1, 3, 5, 8 hours) and Days 2 (24 hours), 3, 4, 5, 6, 7, 8, 15, 22, 29, 50
  Apparent volume of distribution in the terminal phase
Bioavailability (F) | Day 1 (0, 1, 3, 5, 8 hours) and Days 2 (24 hours), 3, 4, 5, 6, 7, 8, 15, 22, 29, 50
  Absolute bioavailability

CONTACTS AND LOCATIONS:
Overall Officials: Libbie McKenzie, MD, Study Director — Veloxis Pharmaceuticals
Locations (1):
- CTI Clinical Research Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No